CLINICAL TRIAL: NCT00099671
Title: A Phase I, Randomized, Placebo-Controlled, Double-Blind Study Evaluating the Safety of Subcutaneous Single Dose Interleukin-7 in HIV-1-Infected Subjects Who Are Receiving Antiretroviral Treatment
Brief Title: Safety of Interleukin-7 in HIV Infected People Currently Taking Anti-HIV Drugs
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A5214; 10022 (Registry Identifier: DAIDS ES Registry Number); ACTG A5214
Record Dates: First submitted 2004-12-17; First posted 2004-12-20 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — Interleukin-7

INTERVENTIONS:
Drug: Recombinant human interleukin-7

SUMMARY:
The purpose of this study is to determine the safety of a single, under-the-skin dose of interleukin-7 (IL-7) in HIV infected people currently taking anti-HIV drugs.

DETAILED DESCRIPTION:
CD4 count is the best predictor of HIV disease progression. IL-7 plays an important role in immune system function, especially in the development of T cells, including CD4 cells. IL-7 may improve HIV-specific immune responses by increasing the number of CD4 cells and boosting immune response. This study will evaluate the safety of a single IL-7 dose given under the skin in HIV infected patients who are currently on potent antiretroviral therapy (ART).

This study will last 13 weeks. Participants will be stratified into two groups by viral load: Stratum 1 participants will have viral loads of less than 50 copies/ml, and Stratum 2 participants will have viral loads between 50 and 50,000 copies/ml. Participants will receive one dose of either IL-7 or placebo at study entry. Five different dosing levels of IL-7 will be tested sequentially in both strata. Dose escalation will occur independently in each stratum and enrollment in a stratum will end when the maximum-tolerated dose is reached. As of 10/23/06, due to adverse events associated with the 60 mcg/kg dose level, all participants will receive up to the 30 mcg/kg dose level, with no further dose escalation. New participants will enroll in Stratum 2 only.

There will be 9 study visits; medical and medication history, a physical exam, lymph node and spleen assessment, and blood collection will occur at most visits. Participants will undergo an electrocardiogram at study entry and on Day 1, and a spleen ultrasound at Week 3. Urine collection will occur on Day 4 and at Weeks 2 and 3.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected
* Currently on ART consisting of at least 3 antiretroviral drugs for at least 12 months prior to study entry and stable (no change in dose) on treatment for at least 3 months prior to study entry
* CD4 count of 100 cells/mm3 or more within 42 days of study entry
* Viral load of 50,000 copies/ml or less within 42 days of study entry
* Willing to use acceptable forms of contraception
* Participants with a Category C AIDS-defining illness during the 12 months prior to study entry may be eligible as long as their CD4 count is 200 cells/mm3 or more at screening. Participants with Kaposi's sarcoma may also be eligible for this study.

Exclusion Criteria:

* Lymphadenopathy greater than 2.0 cm
* Known allergy or sensitivity to study drug or its formulations
* Current drug or alcohol abuse
* Serious illness or hospitalization that, in the opinion of the site investigator, may interfere with the study results
* Prior use of any interleukins
* Systemic cancer chemotherapy, systemic investigational agents, or immunomodulators (e.g., growth factors, systemic corticosteroids, HIV vaccines, immune globulin, interferons) within 90 days prior to study entry
* Heparin within 96 hours prior to study entry, or anticipating the need for heparin within 96 hours after the study injection
* History of cancer (except basal carcinoma of the skin or Kaposi's sarcoma)
* Enlargement of spleen
* History of hypercoagulability (deep vein thrombosis or pulmonary embolism)
* History of seizure disorder
* History of extensive psoriasis, Crohn's disease, uveitis, or other autoimmune disease having induced severe complications
* Significant psychiatric, cardiac, pulmonary, thyroid, renal, or neurological disease requiring therapy
* Positive hepatitis B surface antigen or positive hepatitis C antibody at screening
* Plan to start new ART within 8 weeks after study entry
* Breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2005-04; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Safety, as assessed by dose-limiting toxicities

SECONDARY OUTCOMES:
Change in IL-7 plasma level from study entry to Day 28
concentrations of recombinant human IL-7 (rhIL-7) at study entry (prior to dose) and at 0.5, 1.0, 1.5, 2.0, 2.5, 4, 8, 12, 24, 48, and 72 hours after dose
T-cell proliferation and activation status
lymphocyte subsets prior to study entry, study entry and on Days 1, 2, 4, 14, and 28
anti-IL-7 antibodies prior to study entry and on Days 28 and 56
HIV-1 viral load at baseline and on Days 1, 4, 14, and 28
nine-color advanced flow cytometry on stored peripheral blood mononuclear cells (PBMCs) at baseline and on Days 4 and 28
effect of age on laboratory outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Irini Sereti, MD, Study Chair — National Institute for Allergy and Infectious Diseases, National Institutes of Health; Michael M. Lederman, MD, Study Chair — Case Western Reserve University, University Hospitals of Cleveland
Locations (5):
- United States (5):
  - Univ. of California Davis Med. Ctr., ACTU, Sacramento, California
  - Univ. of Miami AIDS CRS, Miami, Florida
  - Rush Univ. Med. Ctr. ACTG CRS, Chicago, Illinois
  - Case CRS, Cleveland, Ohio
  - MetroHealth CRS, Cleveland, Ohio

REFERENCES:
- [Background] Fry TJ, Mackall CL. Interleukin-7: master regulator of peripheral T-cell homeostasis? Trends Immunol. 2001 Oct;22(10):564-71. doi: 10.1016/s1471-4906(01)02028-2. PMID 11574281
- [Background] Geiselhart LA, Humphries CA, Gregorio TA, Mou S, Subleski J, Komschlies KL. IL-7 administration alters the CD4:CD8 ratio, increases T cell numbers, and increases T cell function in the absence of activation. J Immunol. 2001 Mar 1;166(5):3019-27. doi: 10.4049/jimmunol.166.5.3019. PMID 11207251
- [Background] Kedzierska K, Crowe SM. Cytokines and HIV-1: interactions and clinical implications. Antivir Chem Chemother. 2001 May;12(3):133-50. doi: 10.1177/095632020101200301. PMID 12959322
- [Background] Pett SL, Kelleher AD. Cytokine therapies in HIV-1 infection: present and future. Expert Rev Anti Infect Ther. 2003 Jun;1(1):83-96. doi: 10.1586/14787210.1.1.83. PMID 15482104
- [Result] Sereti I, Dunham RM, Spritzler J, Aga E, Proschan MA, Medvik K, Battaglia CA, Landay AL, Pahwa S, Fischl MA, Asmuth DM, Tenorio AR, Altman JD, Fox L, Moir S, Malaspina A, Morre M, Buffet R, Silvestri G, Lederman MM; ACTG 5214 Study Team. IL-7 administration drives T cell-cycle entry and expansion in HIV-1 infection. Blood. 2009 Jun 18;113(25):6304-14. doi: 10.1182/blood-2008-10-186601. Epub 2009 Apr 20. PMID 19380868
- [Derived] Vandergeeten C, Fromentin R, DaFonseca S, Lawani MB, Sereti I, Lederman MM, Ramgopal M, Routy JP, Sekaly RP, Chomont N. Interleukin-7 promotes HIV persistence during antiretroviral therapy. Blood. 2013 May 23;121(21):4321-9. doi: 10.1182/blood-2012-11-465625. Epub 2013 Apr 15. PMID 23589672